CLINICAL TRIAL: NCT01838993
Title: The Effect of Ultrasonic Nebulizer Delivered Lidocaine on Circulatory Responses During Tracheal Intubation and Postoperative Sore Throat
Brief Title: Inhalation of Lidocaine Before Intubation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: New Taipei City Hospital (Other)
Responsible Party: Principal Investigator, Chen Yen-Po, Physician, New Taipei City Hospital
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CS 2013011
Record Dates: First submitted 2013-04-21; First posted 2013-04-24 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Sore Throat
Keywords: anesthetics,; local,; lidocaine;; nebulizers and vaporizers;; complications,; intubation,; intratracheal.
MeSH Terms: conditions — Pharyngitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lidocaine (Active Comparator): Inhalation of lidocaine before intubation
  Interventions: Drug: Lidocaine inhalation
- Control (Placebo Comparator): Normal saline inhalation before intubation
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lidocaine inhalation — Lidocaine inhalation before intubation
  Arms: Lidocaine
Drug: Placebo
  Arms: Control

SUMMARY:
We investigate the potential benefits of ultrasound-driven lidocaine inhalation immediately before induction.

DETAILED DESCRIPTION:
Sudden increases in blood pressure and heart rate after tracheal intubation and post-operative sore throat are two common undesirable side effects of general anesthesia and might lead to patients' morbidity or dissatisfaction. We investigated the possibility to attenuate both side effects with one single method, i.e. ultrasound-driven lidocaine inhalation immediately before induction.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I or II. Patients scheduled for elective surgery under general anesthesia with orotracheal intubation

Exclusion Criteria:

* patient's refusal to join, major surgery or expected operation duration longer than 3 hours, patients with a anticipated difficult airway, requiring a nasogastric tube in peri-operative stage, having recent upper respiratory tract infection (within 1 week) or pre-existing sore throat.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | 3 min
  Non invasive blood pressure every min for 3 min

SECONDARY OUTCOMES:
Post operative sore throat | 3 days
  Questionnaire for Post operative sore throat

CONTACTS AND LOCATIONS:
Overall Officials: Chen Yen Po, MD, Principal Investigator — New Taipei City Hospital
Locations (1):
- New Taipei City Hospital, New Taipei City, Taiwan